CLINICAL TRIAL: NCT05839561
Title: Management of Tubal Pregnancy With Off-label Use of Letrozole in Monotherapy
Brief Title: Monotherapy With Letrozole in Tubal Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, M.D., Ph.D., Principal Investigator, Jagiellonian University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1072.6120.321.2020
Record Dates: First submitted 2023-04-15; First posted 2023-05-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Tubal Pregnancy Unruptured
Keywords: Tubal pregnancy; Methotrexate; Letrozole
MeSH Terms: conditions — Pregnancy, Tubal | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tubal pregnancy treated with MTX (Active Comparator): MTX in a single dose of 100 mg intravenously on day 0
  Interventions: Drug: MTX as monotherapy
- Tubal pregnancy treated with letrozole (Active Comparator): Letrozole in a daily dose of 5 mg (2 x 2.5 mg) orally for 10 days from day 0
  Interventions: Drug: Letrozole as monotherapy

INTERVENTIONS:
Drug: Letrozole as monotherapy — Letrozole 5 mg daily orally for 10 days from day 0
  Arms: Tubal pregnancy treated with letrozole
Drug: MTX as monotherapy — MTX in a single dose of 100 mg intravenously on day 0
  Arms: Tubal pregnancy treated with MTX

SUMMARY:
It is hypothesized that the inhibition of estradiol production by letrozole may interfere with physiological effects of progesterone necessary to maintain the pregnancy. Treatment of tubal pregnancy with letrozole would allow to avoid the adverse effects of methotrexate (MTX) in women refusing surgery. The aim was to compare the effectiveness of letrozole with MTX in the management of tubal pregnancy.

DETAILED DESCRIPTION:
A prospective cohort study is conducted among women with tubal pregnancy. Women with increasing B-human chorionic gonadotropin (B-hCG) concentrations are included.

Two study arms were planned:

i) women treated with MTX: MTX in a single dose of 100 mg intravenously on day 0; ii) women treated with letrozole: letrozole at a daily dose of 5 mg orally for 10 days from day 0.

The inclusion criteria included B-hCG concentration up to 3000 mIU/ml and no contraindications to conservative treatment. Women who did not meet criteria for conservative treatment were excluded. Blood parameters (B-hCG, hemoglobin, creatinine, urea, alanine/aspartate transaminase, gamma-glutamyltransferase, bilirubin) were tested on days 0,4,7. Cases of treatment failure were counted, i.e. the need to perform laparoscopy due to tubal pregnancy rupture, pain, increase in B-hCG concentration.

The women were given the option to choose the treatment used in the study. All enrolled women gave informed written consent to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* tubal pregnancy confirmed on pelvic ultrasound
* increasing serum B-hCG concentrations in at least two subsequent measures
* serum B-hCG concentration ≤ 3000 mIU/ml

Exclusion Criteria:

* free fluid in lesser pelvis on pelvic ultrasound
* positive fetal heartbeat on pelvic ultrasound
* abdominal pain
* heterotopic pregnancy
* contraindications to MTX

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The effectiveness of the treatment | up to 6 months
  Conversion rate to laparoscopy due to tubal rupture, pain, serum B-hCG increase in the course of treatment

SECONDARY OUTCOMES:
The effect of treatment on bone marrow function (hemoglobin) | up to 6 months
  Changes in hemoglobin concentration (g/dl) in the course of treatment (day 0,4,7)
The effect of treatment on bone marrow function (red blood cells) | up to 6 months
  Changes in red blood cell count (T/l) in the course of treatment (day 0,4,7)
The effect of treatment on bone marrow function (white blood cells) | up to 6 months
  Changes in white blood count (G/l) in the course of treatment (day 0,4,7)
The effect of treatment on bone marrow function (platelets) | up to 6 months
  Changes in platelet count (G/l) in the course of treatment (day 0,4,7)
The effect of treatment on liver function (total bilirubin) | up to 6 months
  Changes in the concentrations of serum total bilirubin (mg/dl) in the course of treatment (day 0,4,7)
The effect of treatment on liver function (alanine transaminase) | up to 6 months
  Changes in the concentrations of alanine transaminase (IU/l) in the course of treatment (day 0,4,7)
The effect of treatment on liver function (aspartate transaminase) | up to 6 months
  Changes in the concentrations of aspartate transaminase (IU/l) in the course of treatment (day 0,4,7)
The effect of treatment on liver function (gamma-glutamyltransferase) | up to 6 months
  Changes in the concentrations of gamma-glutamyltransferase (IU/l) in the course of treatment (day 0,4,7)
The effect of treatment on kidney function (urea) | up to 6 months
  Changes in the concentrations of serum urea (mmol/l) in the course of treatment (day 0,4,7)
The effect of treatment on kidney function (creatinine) | up to 6 months
  Changes in the concentrations of serum creatinine (mg/dl) in the course of treatment (day 0,4,7)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jach, Prof., Ph.D., Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Department of Gynecology and Obstetrics, Clinic of Gynecological Endocrinology, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No